CLINICAL TRIAL: NCT02067780
Title: Evaluation of Two Strategies of Antibiotic Treatment With Levofloxacin in Acute Exacerbation of Chronic Obstructive Pulmonary Disease: Short Treatment-versus Treatment Guided by Markers of Inflammation
Brief Title: Short Antibiotic Treatment Versus Duration Guided by Markers of Inflammation in the Treatment of AECOPD
Acronym: AECOPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COPD levofloxacine Study
Record Dates: First submitted 2014-02-11; First posted 2014-02-20 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention (CRP-guided) group (Experimental): 500 mg (one tablet) of oral levofloxacin daily of levofloxacin for 7 days unless the serum CRP decrease by at least 50% from baseline value. Measurements of serum CRP were done at ED admission, at day-2, day-4 and day-6 and made available to the attending physicians.
  Interventions: Drug: Levofloxacin 500mg
- The standard care (control) group (Experimental): 500 mg of levofloxacin per day for the first two days. Thereafter, oral tablet of placebo was prescribed according to CRP values as in CRP guided group to keep the blindness of the study.
  Interventions: Drug: Levofloxacin 500mg

INTERVENTIONS:
Drug: Levofloxacin 500mg — One tablet per day for 7days.
  Other Names: Placebo Levofloxacin 500mg

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is one of the most common diseases in the world. In a recent study, we showed that administration of levofloxacin is superior to placebo in the treatment of decompensation of COPD; it is accompanied by a substantial reduction in mortality and a significant reduction in the residence time in hospital.

In Tunisia, few data are available on the epidemiology of COPD decompensation. The choice of antibiotic to be used in this situation is challenging to the clinician who must choose between traditional antibiotics (cyclins, aminopenicillins, cotrimoxazole...) and new antimicrobial agents. Recently, it has been emphasized the selection of patients for treatment according to the degree of systemic inflammation (C-Reactive Protein). Indeed, there would have a correlation between the tracheobronchial infection and elevated inflammatory markers. As the elevation of these markers is proportional to the intensity of the inflammatory reaction of the body, is based on the kinetics of these biomarkers in antibiotic treatment seems logical. Thus, C-Reactive Protein allowed not only knowing when to start antibiotics, but also through their kinetic, these markers can guide the duration of therapy and shorten the duration of antibiotic therapy: a rate cut would ensure that the antibiotic treatment was adopted. Available guidelines stated that antibiotic treatment should be maintained at an average of 7 to 10 days while some studies showed no clinical inferiority of courses as short as 3 days. Further reduction of the duration of antibiotherapy was even suggested in order to reduce the risk of adverse events and the pressure that drives bacterial resistance. Hence, we conducted this study using an algorithm to comprehensively evaluate the role of CRP-guided antibiotic prescription in optimizing treatment duration in AECOPD.

DETAILED DESCRIPTION:
This study is a prospective, randomized, double blind controlled study including patients admitted to the emergency department (ED) with AECOPD. Patients were randomly assigned (1:1) to receive treatment either according to guidance based on serum CRP level (CRP-guided group) or the standard of care (control group). The randomisation sequence was generated using the sealed envelope sequence generator stratified according to investigator site. Online inclusion of patients according to the concealed sequence was done with an independent, centralised web-based system (DACIMA Tunisia; https://www.dacimasoftware.com).

Patients were assigned to one of the two treatment arms:

1. the intervention (CRP-guided) group: 500 mg (one tablet) of oral levofloxacin daily of levofloxacin for 7 days unless the serum CRP decrease by at least 50% from baseline value. Measurements of serum CRP were done at ED admission, at day-2, day-4 and day-6 and made available to the attending physicians.
2. the standard care (control) group: 500 mg of levofloxacin per day for the first two days. Thereafter, oral tablet of placebo was prescribed according to CRP values as in CRP guided group to keep the blindness of the study. Also, in order to ensure blinding, active drug as well as placebo tablets were encapsulated for identical appearance and placed in sealed envelopes.

The study is approved by ethics committees of all participating centers prior to implementation, and all included patients provided their written informed consent. The study was. The study protocol has been prepared in accordance with the revised Helsinki Declaration for Biomedical Research Involving Human Subjects and Guidelines for Good Clinical Practice.

After verification of inclusion and exclusion criteria as well the informed consent, demographic, clinical and biological data were collected at baseline. These included patient comorbidities, number of exacerbations in the past year, physical examination findings, blood gas analysis, and standard laboratory tests results. Expectorated sputum samples were collected for pathogen culture. All data were recorded in standardized electronic case report forms. All statistical analyses were performed using SPSS software, version 20.0.

ELIGIBILITY:
Inclusion Criteria:

* patients having COPD (according to the definition of the American Thoracic Society) in acute exacerbation

Exclusion Criteria:

* clinical evidence of hemodynamic compromise with the need for vasoactive drugs
* immediate need for mechanical ventilation,
* Glasgow Coma scale <12,
* pneumonia,
* previous adverse reactions to the study drug,
* antibiotic treatment in the previous days,
* pregnancy or lactation,
* severe renal (creatinine clearance 40 mL/min) or hepatic impairment,
* lung disease other than COPD that could affect the clinical evaluation of the treatments. --active alcohol or drug abuse

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
cure rate | 1 year after starting protocol
  By hospital Data and telephonic calling.

SECONDARY OUTCOMES:
Rate of additional antibiotherapy course | one week
  The frequency of additional antibiotherapy course indicated to treat COPD patients during the hospital stay.
rate of admission in the intensive care unit | one week
  By hospital Data and telephonic calling.
exacerbation rate | 1 year after starting protocol
  By hospital Data and telephonic calling.
exacerbation free interval | 1year after starting protocol
  rate of admission in the intensive care unit

CONTACTS AND LOCATIONS:
Overall Officials: Semir Nouira, professor, Study Director — Research Laboratory (LR12SP18) University of Monastir 5000 Tunisia
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: officiel site — http://www.urgencemonastir.com